CLINICAL TRIAL: NCT04543695
Title: A Prospective, Multicenter, Randomized Controlled Trial of Neoadjuvant Therapy for High-risk Locally Advanced Rectal Cancer
Brief Title: A Study of Total Neoadjuvant Therapy for High-risk Locally Advanced Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Peking Union Medical College Hospital (Other); Jilin Provincial Tumor Hospital (Other); Cancer Hospital of Guizhou Province (Other); Xijing Hospital (Other)
Responsible Party: Principal Investigator, JIN JING, Clinical Professor，Radiotherapy Department, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC201809007
Record Dates: First submitted 2020-08-03; First posted 2020-09-10 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Radiotherapy; High Risk; Total Neoadjuvant Therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy; XELOX

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- adjuvant chemotherapy group (Active Comparator): concurrent chemoradiotherapy → TME → adjuvant chemotherapy (control group)
  Interventions: Combination Product: Concurrent Chemoradiotherapy; Drug: XELOX; Drug: mFOLFOX; Procedure: TME
- consolidation chemotherapy group (CNCT group) (Experimental): concurrent chemoradiotherapy → consolidation chemotherapy → TME (CNCT group)
  Interventions: Combination Product: Concurrent Chemoradiotherapy; Drug: XELOX; Drug: mFOLFOX; Procedure: TME
- induction chemotherapy group (INCT group) (Experimental): induction chemotherapy → concurrent chemoradiotherapy →TME ( INCT group).
  Interventions: Combination Product: Concurrent Chemoradiotherapy; Drug: XELOX; Drug: mFOLFOX; Procedure: TME

INTERVENTIONS:
Combination Product: Concurrent Chemoradiotherapy — Radiotherapy:
  50Gy in 25 fractions to the primary tumor and to mesorectal, presacral,and internal iliac lymph nodes.
  Concurrent chemotherapy:
  Capecitabine 1650 mg/m2/d
Drug: XELOX — Intravenous infusion of oxaliplatin (130 mg/m2 over 2 h) on day 1 and oral administration of capecitabine (1000 mg/m2 twice daily) from day 1 to day 14, is repeated every 3 weeks for 6 cycles.
  6 courses，3 weeks per course
  Other Names: CAOPX
Drug: mFOLFOX — Administration of l-LV (400 mg/m2) and oxaliplatin (85 mg/ m2) by intravenous infusion over 2 h, followed by rapid intravenous infusion (iv) of 5-FU (400 mg/m2) and then slow infusion (civ) of 5-FU (2400 mg/m2 over 46 h), is repeated every 2 weeks for 9 cycles.
Procedure: TME — Total mesorectal excision

SUMMARY:
A Phase II Study of Total Neoadjuvant Therapy for High-risk Locally Advanced Rectal Cancer

DETAILED DESCRIPTION:
Recommended treatment of patients with locally advanced rectal cancer (LARC) includes preoperative chemoradiation (CRT), total mesorectal excision (TME) and postoperative adjuvant chemotherapy (ACT). However, treatments fail to show an improved therapeutic effect on high-risk patients now. Total neoadjuvant therapy (TNT) is a new try for rectal cancer treatment,and this trial aims to identify and select the more promising TNT sequence.

This trail is a multicenter, randomized, phase II trial . Eligible patients age from 18 to 75 years with histologically confirmed rectal adenocarcinoma. MRI is mandatory, and patients of stage II or III rectal cancer are eligible if any of the following criteria are fulﬁlled: Categories T4,Categories N2, MRF involvement, EMVI positive, and lateral lymph node involvement. Patients are randomly assigned to 3 groups, group 1: concurrent chemoradiotherapy → TME → adjuvant chemotherapy (control group);or group 2: concurrent chemoradiotherapy → consolidation chemotherapy → TME (CNCT group);Or group 3: induction chemotherapy → concurrent chemoradiotherapy →TME ( INCT group).The primary end point is the rate of tumor down-staging, which is deﬁned as stage yp0-II after surgery,and watch-and-wait strategy after complete clinical response (cCR) was allowed. Secondary end points include acute toxicity, compliance with TNT, surgical complications, 3-year overall survival (3yOS),3-year disease free survival (3yDFS),3-year distant metastatic free survival(3yDMFS),3-year locoregional recurrence-free survival(3yLRRFS) and quality of life.

ELIGIBILITY:
Inclusion criteria:

1. 18-75 years old, regardless of gender
2. Histologically confirmed rectal adenocarcinoma;
3. Up to 12 cm above the anal verge on the basis of rigid rectoscopy.
4. MRI of the rectum is acceptable;
5. Patients in stage II or III rectal cancer are eligible if any of the following criteria are fulﬁlled: Categories T4,Categories N2, MRF involvement, EMVI positive, and lateral lymph node involvement.
6. ECOG score 0-1 or KPS score ≥80.

Exclusion Criteria:

1. History of malignant tumor in other parts;
2. Cannot complete MRI; Allergic to 5-fu drugs; Allergic to platinum drugs;
3. During thrombolytic and anticoagulant therapy, the patient has bleeding diathesis or coagulation dysfunction; Or aneurysm, stroke, transient ischemic attack, arteriovenous malformation in the past year;
4. History of kidney, urine test found proteinuria or clinical renal function was significantly abnormal;
5. History of digestive tract fistula, perforation or severe ulcer;
6. Active infection is present; Clinically obvious heart disease; New York heart association (NYHA) of Ⅱ level or congestive heart failure; Unstable symptomatic arrhythmia or peripheral vascular disease ≥ grade II; Myocardial infarction and cerebrovascular accident occurred within 6 months before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The rate of tumor down-staging | 6-8 months
  Tumor down-staging is considered as Stage yp0-II after surgery, and watch-and-wait strategy after complete clinical response (cCR) was allowed.

SECONDARY OUTCOMES:
Rate of compliance with TNT | 6-8 months
  Rate of compliance with TNT
3y OS | 3years
  3-year overall survival (3yOS)
3y DFS | 3years
  3-year disease free survival (3yDFS)
3y DMFS | 3 years
  3-year distant metastatic free survival(3yDMFS)
3y LRRFS | 3 years
  3-year locoregional recurrence-free survival(3yLRRFS)
EORTC QLQ-C30 | 3 years
  EORTC QLQ-C30 to assess the quality of life
EORTC QLQ-CR29 | 3 years
  EORTC QLQ-CR29 to assess the quality of life
Wexner continence grading scale | 3 years
  Wexner continence grading scale
CTCAE 4.0 | 6-8months
  Severe acute adverse reaction rate（≥III degree）
Incidence of surgical complications | 6-8 months
  Incidence of surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, M.D., Study Director — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No